CLINICAL TRIAL: NCT06082440
Title: A Single-Arm Clinical Study on the Safety and Tolerance of Human Umbilical Cord Mesenchymal Stem Cells Mediated by Arthroscopy in Patients With Stage II-III Knee Osteoarthritis
Brief Title: Study on the Safety and Tolerance of Mesenchymal Stem Cells Mediated by Arthroscopy in Patients With Osteoarthritis
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Wannan Medical College (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QWang
Record Dates: First submitted 2023-09-25; First posted 2023-10-13 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2023-10

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Human Umbilical Mesenchymal Stem Cells (Experimental): Participants received a single administration for Human Umbilical Mesenchymal Stem Cells during the treatment period.The specification is 2.5 × 10^7cells/2ml suspension/branch.
  Interventions: Biological: Human Umbilical Mesenchymal Stem Cells

INTERVENTIONS:
Biological: Human Umbilical Mesenchymal Stem Cells — Ntra-articular injection inject a corresponding dose of cells suspension into each joint cavity according to the lesion site.

SUMMARY:
The goal of this clinical trial is to evaluate the safety and tolerability of human umbilical cord mesenchymal stem cells mediated by arthroscopy in patients with knee osteoarthritis. This experiment proposes to enroll 18-22 patients. The experimental drug is human umbilical cord mesenchymal stem cells.

DETAILED DESCRIPTION:
This study adopts a design for a single-dose increasing, single-center, randomized, placebo-controlled trial to explore the safety, tolerance and preliminary efficacy of the single-dose administration of human umbilical cord mesenchymal stem cells mediated by arthroscopy in patients with knee osteoarthritis, as well as to provide a basis for the subsequent clinical study of drug delivery plans.

The experimental process of this study is divided into four stages: screening period, baseline period, study treatment and safety observation period, follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Age range from 40 to 60 years old (including threshold), regardless of gender；
2. According to the 《Chinese Guidelines for the Diagnosis and Treatment of Osteoarthritis (2021 Edition)》, patients diagnosed with knee osteoarthritis；
3. According to the imaging examination results (knee joint X-ray anterolateral axial position), the target knee joint with Kellgren Lawrence grading is classified as Grade II-III；
4. WOMAC pain sub item with a score of at least 4 points and pain lasting for at least 4 weeks from the time of signing the informed consent form；
5. Pain persists for more than six months, or after routine clinical treatment, such as hormone, opioid drugs, viscoelastic supplement therapy, etc., osteoarthritis relapses or worsens again after discontinuation of medication；
6. Those who have continuously used non-steroidal anti-inflammatory drugs for at least 12 weeks and have stabilized their dosage for at least 4 weeks before the first administration, and have maintained a stable medication regimen within 4 weeks after cell therapy；
7. All subjects and their partners who have no family planning within 6 months from screening to the end of the trial and agree to take effective non drug contraceptive measures during the trial period；
8. Those who voluntarily participate in clinical research, understand and sign an informed consent form.

Exclusion Criteria:

1. Those who receive physical therapy of knee joint (bilateral or either side) or use traditional Chinese patent medicines and simple preparations to treat knee arthritis (bilateral or either side) within 6 weeks before treatment；
2. Within 3 months before the start of treatment, patients who have received topical glucocorticoid therapy on both sides or either side of the knee joint, or have received systemic glucocorticoid therapy, or who require systemic glucocorticoid therapy during the study period；
3. Individuals who have undergone knee arthroscopic surgery or other open surgeries related to knee joint operations within the first 6 months of the screening period；
4. Individuals who have received any medication injection treatment within the knee joint (bilateral or either side) cavity within 6 months before the start of treatment；
5. Patients who have received opioid therapy for knee osteoarthritis 4 weeks before the start of treatment；
6. Those who have undergone or need to undergo knee replacement surgery during the trial period；
7. Diagnosed as secondary knee osteoarthritis；
8. Patients with knee joint damage caused by other reasons, or inflammatory and painful diseases that affect the knee joint or affect the joint；
9. Other lower limb diseases that may interfere with the evaluation of knee joint efficacy, such as fibromyalgia, obvious back pain, lumbar disc herniation, etc；
10. Patients with skin disorders at the intended injection site of the target knee joint；
11. Individuals with severe systemic or local knee joint infections within the first 3 months of the screening period；
12. Individuals with solid tumors within 5 years prior to screening；
13. Individuals with severe and poorly controlled concomitant diseases；
14. Severe heart disease patients (NYHA heart function level III and above)；
15. Individuals with a clear history of mental disorders, or a history of abuse of psychotropic substances or drug use；
16. Individuals who may be allergic to any component or albumin in experimental biological products.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Estimated)
Dates: Start 2023-11-22 (Actual); Primary Completion 2025-08-15 (Estimated); Study Completion 2026-01-10 (Estimated)

PRIMARY OUTCOMES:
Within 4 weeks after treatment, evaluate the incidence and severity of adverse events. | Within 4 weeks after treatment
  According to the NCI CTCAE v5.0 grading standard, adverse events in the study will be described and the level of them assessed. Then it will be counted up that the number and incidence of drug-related adverse events/adverse reactions, serious adverse events/serious adverse reactions (level 3 or above), and adverse events/adverse reactions leading to withdrawal in each group during the treatment period.
Within 4 weeks after treatment, evaluate the Maximum Tolerable Dose (MTD). | Within 4 weeks after treatment
  The degree of adverse events observed in the experiment will be determined according to the NCI CTCAE v5.0 grading standard. If there were drug-related adverse events of level 3 or above that occurred in half or more of the subjects in any dose group before the dose was reached 1.0 × 10^8 cells/person/time, the dose ramp would be terminated and then the previous dose would be defined as MTD. If not, define 1.0 × 10^8 cells/person/time as MTD.

SECONDARY OUTCOMES:
Evaluate changes on the scores of the Western Ontario and McMaster Universities Osteoarthritis Index relative to baseline after treatment | Baseline, Week 4, Week 12, Week 24 and Week 48
  In the Western Ontario and McMaster Universities Osteoarthritis Index, the minimum value is 0 and the maximum value is 96, and higher scores mean a worse outcome.
Evaluate changes on the degree of the Kellgren-Lawrence grading standard for Knee joint X-ray relative to baseline after treatment | Baseline, Week 24 and Week 48
  In the Kellgren-Lawrence grading standard for Knee joint X-ray, the lowest class is 0 and the highest class is IV, and higher grade means a worse outcome.
Evaluate changes on the degree of the Kellgren-Lawrence grading standard for Knee joint MRI relative to baseline after treatment | Baseline, Week 24 and Week 48
  In the Kellgren-Lawrence grading standard for Knee joint MRI, the lowest class is 0 and the highest class is IV, and higher grade means a worse outcome.
Evaluate changes on the level of inflammatory factors relative to baseline after treatment | Baseline, Week 4, Week 12, Week 24 and Week 48
  At various time frame (baseline, week 4, week 12, week 24 and week 48), it will be measured that the levels of inflammatory factors (IL-1, IL-6, tumor necrosis factor α, PEG2) in the knee joint cavity. Then the changes on the level of inflammatory factors from baseline after treatment will be assessed.
Evaluate changes on the scores of the Visual Analogue Scale relative to baseline after treatment | Baseline, Week 4, Week 12, Week 24 and Week 48
  In the Visual Analogue Scale, the minimum value is 0 and the maximum value is 10, and higher scores mean a worse outcome.
Evaluate changes on the scores of the 36-Item Short Form Survey relative to baseline after treatment | Baseline, Week 4, Week 12, Week 24 and Week 48
  In the 36-Item Short Form Survey, the minimum value is 0 and the maximum value is 900, and higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Qiang Wang, Principal Investigator — First Affiliated Hospital of Wannan Medical College
Locations (1):
- First Affiliated Hospital of Wannan Medical College, Wuhu, Anhui, China

IPD SHARING:
Plan to Share IPD: No